CLINICAL TRIAL: NCT01530568
Title: A Randomised Control Trial of a Standardised and User-friendly Real-time PCR Assay for the Diagnosis of TB Using Tracheal Aspirates Obtained From Patients in the ICU
Brief Title: Gene Xpert Diagnosis of TB Using Tracheal Aspirates From Intensive Care Unit (ICU) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Keertan Dheda, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TB Xpert ICU
Record Dates: First submitted 2012-01-24; First posted 2012-02-10 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Tuberculosis
Keywords: Intensive care, TB, tracheal aspirates, Gene Xpert
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smear (Active Comparator): Routine microbiology based diagnostics for TB
  Interventions: Other: Smear
- GeneXpert (Experimental): Arm that will receive the Xpert test
  Interventions: Other: Xpert

INTERVENTIONS:
Other: Xpert — This arm receives the GeneXpert test
  Arms: GeneXpert
Other: Smear — This arm receives smear microscopy
  Arms: Smear

SUMMARY:
Aim:

To evaluate the diagnostic utility and impact on patient outcomes of an automated PCR (Gene Xpert® MTB/RIF), in a group of patients with suspected pulmonary TB who are mechanically ventilated in ICU, using tracheal aspirates.

Hypothesis:

Gene Xpert is an accurate tool for the diagnosis of TB in the Intensive Care Unit and will impact on rates of treatment initiation and hospital stay.

DETAILED DESCRIPTION:
Background Tuberculosis (TB) is a serious global public health emergency and there is a great need for the improvement of current diagnostic tools and the evaluation of newer and novel technologies for the rapid diagnosis of TB. The most common testing method for TB is sputum smear microscopy, which has remained largely unchanged in its sophistication and sensitivity. Smear microscopy detects around 50% of all active TB cases and is not capable of identifying drug resistance. Furthermore, even though culture is more accurate results are only available in several weeks. Treating patients empirically for TB exposes patients to the toxic side-effects of drugs, and if there is no response to treatment, raises the question of MDR-TB. These considerations apply to clinical decision-making in the ICU where TB is not infrequently encountered. A diagnosis of TB in this setting has important implications for drug-drug interactions, route of administration, and drug toxicity.

The Gene Xpert® system's MTB/RIF Assay, an on-demand molecular test for simultaneous detection of Mycobacterium tuberculosis (M.tb) and rifampicin (RIF) resistance, has recently been released. This is the only system that combines on-board sample preparation with real-time PCR [1]. Helb and colleagues developed and performed the first analysis of the Cepheid Gene Xpert System's MTB/RIF assay. They evaluated the diagnostic utility of the system using sputum samples and showed that the system was highly sensitive and simple-to-use [2]. A recent paper (NEJM, 2010, in press) that enrolled almost 2000 patients found Xpert to have a sensitivity of almost 90% in smear-negative TB. However, how the test will perform when using tracheal aspirates is unknown. It is also unclear whether the test will have any impact in the ICU where the decision to treat is often made clinically and empiric treatment is initiated. To address these questions we aim to obtain tracheal aspirates from about 120 mechanically ventilated patients with suspected TB from the Groote Schuur Hospital Intensive Care Unit. Tests will be conducted at the Lung Infection and Immunity Unit laboratory (Groote Schuur Hospital, Cape Town) to evaluate the diagnostic utility of the Xpert® MTB/RIF Assay in this group of patients. The expected study period will be 12 months.

ELIGIBILITY:
Inclusion criteria:

1. Any ventilated patients over 18 years of age with suspected TB (suggestive pulmonary infiltrates, a history of constitutional symptoms preceding the ICU admission, or patients known or suspected to be infected with the human immunodeficiency virus (HIV)).

Exclusion criteria:

1. Patients known to have active TB or to already be on antituberculous medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Rates of TB treatment initiation | 48 hours
  The proportion of patients on TB treatment in each arm will be compared longitudinally

SECONDARY OUTCOMES:
Mortality in ICU | up to 2 months
  The time-specific proportion of patients who have died prior to discharge will be compared across arms
Duration of mechanical ventilation | Up to 2 weeks
  The median Duration of mechanical ventilation will be compared between arms prior to discharge up to 2 weeks
ICU length of stay | up to 3 months
  The median ICU length of stay will be compared up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, which operates within the Cape Town Central Health District of the Metro Region, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Calligaro GL, Theron G, Khalfey H, Peter J, Meldau R, Matinyenya B, Davids M, Smith L, Pooran A, Lesosky M, Esmail A, Miller MG, Piercy J, Michell L, Dawson R, Raine RI, Joubert I, Dheda K. Burden of tuberculosis in intensive care units in Cape Town, South Africa, and assessment of the accuracy and effect on patient outcomes of the Xpert MTB/RIF test on tracheal aspirate samples for diagnosis of pulmonary tuberculosis: a prospective burden of disease study with a nested randomised controlled trial. Lancet Respir Med. 2015 Aug;3(8):621-30. doi: 10.1016/S2213-2600(15)00198-8. Epub 2015 Jul 22. PMID 26208996